CLINICAL TRIAL: NCT03008434
Title: Traumatic Brain Injury and Yoga
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Arlene Schmid, Principal Investigator, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-5905H
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Brain Injury
Keywords: yoga; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga Group (Experimental): Yoga twice a week for 8 weeks focusing on balance and pain.
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Yoga Group: designed for chronic TBI was provided two times a week for 8 weeks.

SUMMARY:
This long-term goal of this project was to advance best practices in occupational therapy in conjunction with yoga. To address the long-term goal, this research team developed a pilot yoga intervention. The intervention was designed to focus on balance, balance confidence, body responsiveness, pain, physical ability and quality of life. Assessments were then chosen to address these areas pre and post yoga intervention. A manual and protocol were developed for the intervention and then the intervention was implemented with a group of individuals with chronic traumatic brain injury.

DETAILED DESCRIPTION:
This was an 8-week yoga intervention, focused on demonstrating the preliminary feasibility and efficacy of yoga for individuals with chronic traumatic brain injury. The study was a mixed-methods longitudinal study. Assessments were conducted 8 weeks prior to the yoga intervention and then just following the 8 week yoga intervention. The objectives of this feasibility and efficacy study was to 1) further develop, standardize, and manualize the yoga for the traumatic brain injury intervention and 2) assess change in balance, balance confidence, body responsiveness, pain, physical ability, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* chronic TBI (>6 months)
* greater than or equal to 18 years of age
* no consistent practice of yoga in the last year

Exclusion Criteria:

* inability to provide informed consent
* less than 18 years of age
* self-report of exercise restriction
* consistent yoga practice within the last year
* inability to attend sessions based on transportation restrictions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 8 weeks
  14 items to assess balance 14 items to assess balance 14 items to assess balance

SECONDARY OUTCOMES:
Activities Balance Confidence Scale | 8 weeks
  Assess balance self-efficacy or confidence to maintain balance while performing different actions.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Schmid, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No